CLINICAL TRIAL: NCT04317911
Title: Catheter Ablation for Atrial Fibrillation in Heart Failure With Preserved Ejection Fraction
Brief Title: Catheter Ablation for Atrial Fibrillation in Preserved Ejection Fraction
Acronym: AFFECT
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Principal Investigator, Maura Zylla, Dr. med., University Hospital Heidelberg
Other Study IDs: UKHD-2-520/2015
Record Dates: First submitted 2020-03-13; First posted 2020-03-23 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation
Keywords: Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Catheter Ablation — Patients with preserved ejection fraction presenting for catheter ablation via of atrial fibrillation are included in this study and prospectively observed regarding arrhythmia-related, functional and biomarker-associated outcomes.

SUMMARY:
Atrial fibrillation (AF) displays high prevalence in heart failure with preserved ejection fraction (HF-PEF) and compromises prognosis of affected patients. This study aims to assess catheter ablation (CA) for AF in patients with HF-PEF compared to AF-patients without systolic or diastolic dysfunction. Primary endpoints are freedom from AF and quality of life at 1 year. Furthermore, the study is designed to elucidate mechanistic characteristics distinguishing arrhythmic substrate and predicting AF-recurrence in patients with HF-PEF. For this purpose, left atrial concentrations of biomarkers for inflammation, fibrosis and neurohumoral activation are determined and hemodynamic measurements are performed periprocedurally.

Information on benefit from CA in these patients is necessary for clinical decision making and mechanistic investigations may point to tailored approaches in order to increase therapeutic efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular ejection fraction ≥50%
* Scheduled for catheter ablation of AF

Exclusion Criteria:

* Significant valvular heart disease
* Coronary artery disease with >70% stenoses or necessary coronary Intervention at time of recruitment
* Coronary intervention 60 days before recruitment
* Coronary bypass surgery 90 days before recruitment
* Cardiomyopathy or cardiac storage disease (e.g. amyloidosis)
* Reduced left ventricular ejection fraction
* Pericardiac disease
* Significant pulmonary hypertension
* Chronic obstructive pulmonary disease with home-oxygen-therapy, oral steroids, hospitalization due to exacerbations during the last 12 months before recruitment, or suspected severe pulmonary condition based on clinical evaluation
* Other non-cardiac conditions associated with limited physical capacity (adipositas permagna, severe anemia)
* Pregnancy
* Other limitations for adequate performance of stress echocardiography (e.g. orthopedic reasons)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting for evaluation for CA of AF with a left ventricular systolic ejection fraction ≥50% are identified and invited to undergo further stratification. All patients are submitted to thorough clinical screening for signs and symptoms of heart failure, echocardiographic assessment of diastolic function and blood test for peripheral plasma levels of natriuretic peptides. Based on these parameters, patients with heart failure with preserved ejection fraction (HF-PEF) are identified according to current guidelines. Patients not meeting HF-PEF-criteria are included in the control group. Their data and follow-up results are gathered in a registry from which age- and gender-matched controls are extracted for comparison with respective matched HF-PEF-cases.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Arrhythmia recurrence | 12 months
  Clinical arrhythmia and holter-recording

SECONDARY OUTCOMES:
nTproBNP | 12 months
  [ng/L]
Troponin T | 12 months
  [pg/mL]
Systolic left ventricular function in echocardiography | 12 months
  LVEF [%]
Diastolic left ventricular function in echocardiography | 12 months
  E/e'
PA-pressure in echocardiography | 12 months
  [mmHg]
Quality of life questionnaire | 12 months
  SF-36
Diastolic function in stressechocardiography | 12 months
  E/e'
6-minute-walk-test | 12 months
  [m]

CONTACTS AND LOCATIONS:
Overall Officials: Maura M Zylla, Dr. med., Principal Investigator — University Hospital Heidelberg, Department of Cardiology (Prof. Dr. H.A. Katus)
Locations (1):
- University Hospital Heidelberg, Department of Cardiology, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zylla MM, Leiner J, Rahm AK, Hoffmann T, Lugenbiel P, Schweizer P, Scholz E, Mereles D, Kronsteiner D, Kieser M, Katus HA, Frey N, Thomas D. Catheter Ablation of Atrial Fibrillation in Patients With Heart Failure and Preserved Ejection Fraction. Circ Heart Fail. 2022 Sep;15(9):e009281. doi: 10.1161/CIRCHEARTFAILURE.121.009281. Epub 2022 Jun 21. PMID 36126143